CLINICAL TRIAL: NCT01544374
Title: Implementing a Tracking & Feedback Registry to Allay Cancer Therapy Disparities
Brief Title: Tracking & Feedback Registry to Reduce Breast Cancer Treatment Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 09-1155; 5R01CA149025 (NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-03-05 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Treatment Disparities; Tracking and Feedback; Registry; Cancer Therapy Disparities; Adjuvant Treatment; Racial Disparities; Underuse of Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tracking & Feedback (Experimental): Systems based intervention tracking oncology consultations and feeding back information to surgeons
  Interventions: Other: Tracking & Feedback
- Control- no intervention (No Intervention): Usual Care

INTERVENTIONS:
Other: Tracking & Feedback — Systems based intervention tracking oncology consultations and feeding back information to surgeons
  Arms: Tracking & Feedback

SUMMARY:
Breast cancer is the second most common cause of cancer death in women. Black women are less likely than white women to develop breast cancer but, they are more likely to die of the disease. Some of this survival discrepancy is likely due to underuse of adjuvant therapies proven to increase survival. Breast cancer treatment often requires coordination among surgeons, pathologists, primary care physicians, medical and radiation oncologists. In NYC, black and Hispanic women who accessed care and underwent surgical treatment of their breast cancer were twice as likely as whites to experience underuse of adjuvant treatment. Disturbingly, 1/3 of these underuse cases were episodes in which the surgeon recommended treatment, the patient did not refuse and yet, care did not ensue. Underuse in such circumstances is attributable to system failures than to specific provider or patient factors.

In this proposed randomized controlled trial, the investigators aim to test the effectiveness of a Tracking and Feedback (T&F) registry innovation to increase rates of completed oncology consultation and reduce both underuse of needed adjuvant therapy and racial disparities in receipt of these treatments. The investigators also aim to assess the feasibility of implementing a T&F Registry in these high-risk hospitals by evaluating implementation effectiveness for that innovation. The investigators have recruited 10 hospitals that serve large proportions of minority women with breast cancer. The investigators will randomize hospitals and aim to recruit 354 women with a new breast cancer, 177 per intervention arm. The investigators choose these "high risk" hospitals because they serve predominantly minority populations, and such hospitals have higher rates of the system failure cause of underuse, and particularly, the type of underuse targeted by our Tracking and Feedback Registry.

DETAILED DESCRIPTION:
Breast cancer is the second most common cause of cancer death in women. Black women are less likely than white women to develop breast cancer but, they are more likely to die of the disease. Some of this survival discrepancy is likely due to underuse of adjuvant therapies proven to increase survival. Breast cancer treatment often requires coordination among surgeons, pathologists, primary care physicians, medical and radiation oncologists. In NYC, black and Hispanic women who accessed care and underwent surgical treatment of their breast cancer were twice as likely as whites to experience underuse of proven-effective adjuvant treatment. Disturbingly, 1/3 of these underuse cases were episodes in which the surgeon recommended treatment, the patient did not refuse and yet, care did not ensue. Underuse in these circumstances was attributed to system failures rather than to provider or patient factors. Such system failures occurred more often among minority women and among women treated at hospitals serving predominantly minority patients. To target these system failures at 6 NYC hospitals, 4 of which served predominantly minority patients, we used a quasi-experimental pre-post test design to implement a tracking and feedback registry. The Tracking and Feedback registry closed the referral loop between surgeons and oncologists, increased the rate of completed oncology consultations, increased treatment rates and eliminated the racial disparity in underuse. Its effects were greatest at the 4 hospitals serving predominantly minority women, sites that had an EMR and patient navigation prior to and during the T&F implementation. However, the trial was not randomized, tracking and feedback functions were performed by study personnel and not embedded in the hospital's workflow and details of what the surgeons did in response to the feedback was not assessed, resulting in a call for more work in this area.

In this proposed randomized controlled trial, we will implement the Tracking and Feedback (T&F) innovation in hospitals serving predominantly minority women. We will test the effectiveness of the Tracking and Feedback registry innovation to increase rates of completed oncology consultation, reduce underuse of needed adjuvant therapy and racial disparities in receipt of these treatments. We will also assess the feasibility of implementing a T&F Registry in these high-risk hospitals by evaluating implementation effectiveness for this innovation. We have recruited 10 hospitals that serve large proportions of minority women with breast cancer. We will randomize hospitals and will recruit 354 women with a new breast cancer, 177 per intervention arm. We choose these "high risk" hospitals because they serve predominantly minority populations, and such hospitals have higher rates of the system failure cause of underuse, specifically, the type of underuse targeted by our Tracking and Feedback Registry. We will: adapt existing laptop-based Tracking & Feedback software to create a protected web-based format easily accessible to all participating hospitals; tailor the Tracking & Feedback registry to each of the participating hospitals' appropriate workflows including the areas of pathology, surgery, medical and radiation oncology and tumor registry personnel in the process; and embed the tracking and feedback tasks within existing hospital structures and personnel to increase likelihood of sustainability beyond the grant. We will include in the web-based T&F Registry an electronic data capture system to assess responses and actions to the tracking information that is fed back to the surgeons. To assess the T&F Registry's effectiveness, we will compare rates of underuse of patients treated at intervention versus control hospitals. To assess implementation effectiveness at each hospital, we will assess process and outcomes using qualitative and quantitative methods. Qualitatively, we will conduct pre- & post-intervention interviews with key stakeholders to assess the implementation climate and stakeholders' views of the Registry's utility. Quantitatively, we will measure and track actions taken in response to the feedback information. As there is variability across hospitals, we will also assess each hospital's treatment rates both pre- (N=540) and post-intervention (N=354) to provide additional quantitative measures of implementation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are English or Spanish speaking, with a new primary stage 1 or 2 and with tumors > 1 cm or < 1 cm and poorly differentiated breast cancer who have undergone either breast conserving surgery or mastectomy at 1 of 10 participating hospitals in the NY Metropolitan Area.
* All surgeons performing breast surgery at study participating hospitals

Exclusion Criteria:

* Patients with a poor prognosis due to end-stage organ failure or other concomitant conditions such as those undergoing treatment for other cancers

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in intervention effect of adjuvant treatment | at baseline and at one year
  We will compare at initiation and completion of adjuvant treatment on all enrolled patients to determine the intervention's effect

SECONDARY OUTCOMES:
Organizational Characteristics | at 5 years
  To describe the organizational characteristics and the implementation climate of the hospitals and their relationship to the hospitals' change in rates of guideline concordant adjuvant treatment pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Bickell, MD, MPH, Principal Investigator — Icahn School of Medicine Mount Sinai
Locations (11):
- United States (11):
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - University Hospital of Brooklyn at Long Island College Hospital, Brooklyn, New York
  - Kings County Hospital, Brooklyn, New York
  - Lutheran Medical Center, Brooklyn, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Hospital Center, Jamaica, New York
  - Metropolitan Hospital Center, New York, New York
  - Bronx-Lebanon Hospital, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Derived] Bickell NA, Shah A, Castaldi M, Lewis T, Sickles A, Arora S, Clarke K, Kemeny M, Srinivasan A, Fei K, Franco R, Parides M, Pappas P, McAlearney AS. Caution Ahead: Research Challenges of a Randomized Controlled Trial Implemented to Improve Breast Cancer Treatment at Safety-Net Hospitals. J Oncol Pract. 2018 Mar;14(3):e158-e167. doi: 10.1200/JOP.2017.026534. Epub 2018 Jan 3. PMID 29298115
- [Derived] Bickell NA, Moss AD, Castaldi M, Shah A, Sickles A, Pappas P, Lewis T, Kemeny M, Arora S, Schleicher L, Fei K, Franco R, McAlearney AS. Organizational Factors Affect Safety-Net Hospitals' Breast Cancer Treatment Rates. Health Serv Res. 2017 Dec;52(6):2137-2155. doi: 10.1111/1475-6773.12605. Epub 2016 Nov 14. PMID 27861833